CLINICAL TRIAL: NCT05144620
Title: 3D Printing for Pre-Surgical Planning
Acronym: 3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-3135.cc
Record Dates: First submitted 2021-09-27; First posted 2021-12-03 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Surgical Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Imaging (Experimental)
  Interventions: Diagnostic Test: 3D Mapping

INTERVENTIONS:
Diagnostic Test: 3D Mapping — 3D model will be made from diagnostic imaging for pre-surgical planning

SUMMARY:
3D printing is emerging as a new diagnostic tool for pre-surgical planning. 3D printed models are extremely advantageous to surgeons in their preoperative planning. Handling these physical replicas engages active spatial perception skills, enabling a more comprehensive understanding of the presented information in an inherently intuitive manner that cannot be achieved with conventional methods of imaging review that use screen based 2D and volume rendered representations. The investigators are developing a novel technique to create 3D models derived directly from extremely high-resolution medical images that are superior in spatial and contrast resolution to current 3D modelling methods. This produces patient specific models that contain previously unachievable special fidelity and soft tissue differentiation.

Investigators hypothesize that the preoperative use of these new diagnostic quality models will reduce surgical time and improve post-surgical outcomes in the near future. This prospective project will optimize the quality of these 3D models to create highly useful pre-surgical models. Investigators will target those subspecialist areas of the multidisciplinary surgical and imaging team where it is believed these models will have the most impact. The proposed prospective study has two major goals: 1) Investigate the use of uncompressed, ultrahigh resolution CT/MR datasets to produce diagnostic 3D models with identical spatial/contrast resolution to the acquired datasets in the target areas of congenital cardiothoracic surgery, neurosurgical tumor resection and nephrectomy. 2) Compare the accuracy of this innovative method for 3D printing to radiological images and pathological data when available.

DETAILED DESCRIPTION:
The tangible outcome of this research will be measured in a comparative study. The investigators will compare the 3D printed models, resulting from the development of this iterative process of generating models from ultra-high resolution medical images and review by all parties, to radiological images and pathological data. The study team will employ non-biased methods to quantify the results of this comparative study. There will be no randomization and all subjects will receive the same treatments and all outcomes are data focused. Models will not be used for patient treatment and will be used only as to aid preparation and will not be used as a therapeutic device. For this reason, the study team will not prospectively consent subjects.

ELIGIBILITY:
Inclusion Criteria:

* - Patients seen at UCHealth/CHCO and NOC sites between 6/1/2021 - 6/1/2026
* Pregnant women and their fetuses

Exclusion Criteria:

* - Patients 65 and older

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Comparing 3D Models as a new diagnostic tool for pre-surgical training to reduce surgical time | 3 years
  Focus on using pre-operative imaging for producing 3D models for 3 specific presurgical evaluations 1) Adult Clear Cell Renal Mass with a focus on partial nephrectomies. 2) Pediatric Cardiothoracic Surgery 3) Pediatric Neurosurgical primary brain tumor resection involving eloquent areas of the brain (eg speech center, auditory center, visual center, motor cortex, and sensory cortex). 4) Plastic Surgery and Craniomaxillofacial disciplines with a focus on DIEP Flap reconstructions and Alveolar Bone Graft procedures.
  Change in surgical time based on using a 3D model per-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Jacobson, Principal Investigator — Colorado Research Center
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Children's Hospital Colorado, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobson NM, Carerra E, Treat A, McDonnell M, Mathes D, Kaoutzanis C. Hybrid modeling techniques for 3D printed deep inferior epigastric perforator flap models. 3D Print Med. 2023 Sep 12;9(1):26. doi: 10.1186/s41205-023-00181-z. PMID 37700101